CLINICAL TRIAL: NCT03632746
Title: Verifying the Specificity of the Method Combining Nomogram and Sentinel Lymph Node in Predicting Lymph Node Metastasis in Early Gastric Cancer Patients: a Prospective, Single Arm, Observational Study
Brief Title: Verifying the Specificity of a New Method in Predicting Lymph Node Metastasis in Early Gastric Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhaode Bu, MD (Other)
Responsible Party: Sponsor-Investigator, Zhaode Bu, MD, Principal Investigator, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Other Study IDs: Pre gastric preserving study
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Early Gastric Cancer; Lymph Node Metastases
MeSH Terms: conditions — Stomach Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early gastric cancer is defined as gastric cancer that only invades mucosal or submucosal layer. The 5-year survival rate of gastric cancer can exceed 90% due to appropriate treatment. The most important consideration is whether there is lymph node metastasis. Preoperative examination including gastroscopy, endoscopic ultrasonography (EUS) and CT are not accurate enough to predict lymph node metastasis in early gastric cancer. In a retrospective study, we created a nomogram to predict lymph node metastasis in early gastric cancer. In prospective validation, the sensitivity and specificity of the nomogram was 75% and 91%, respectively. Sentinel lymph node is a promising concept in early gastric cancer. Using carbon nanoparticles as tracer, the sensitivity and specificity of sentinel lymph node predicting lymph node metastasis in early gastric cancer were 90% and 100%. Based on these results, we proposed a new method that combines the Nomogram and sentinel lymph node to predict lymph node metastasis in early gastric cancer. First, the probability of lymph node metastasis of early gastric cancer patients is calculated by the Nomogram. Those with low incidence of lymph node metastasis continue to the sentinel lymph node procedure. A patient will be considered non lymph node metastasis if his/her frozen pathology of the sentinel lymph nodes is negative during the surgery. Then the standard radical gastrectomy is performed with lymphadenectomy. By comparing postoperative pathology and sentinel lymph node frozen pathology, the specificity of Nomogram combining sentinel lymph node predicting lymph node metastasis in early gastric patients is calculated. The primary endpoint of this research is that the specificity of the above-mentioned method is over 95%.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as gastric cancer by gastroscopy
* pathologically confirmed as adenocarcinoma
* ages between 18 and 80
* gastroscopy, abdominal enhanced CT and EUS completed
* clinical stage T1N0M0
* the score of the Nomogram less than 110
* potential resectable gastric cancer
* signed informed consent

Exclusion Criteria:

* absolute indication for endoscopic submucosal dissection (ESD)
* tumor located in esophagogastric junction (EGJ)
* accepted adjuvant therap
* pregnant or breast feeding
* history of upper abdominal surgery (laparoscopic cholecystectomy not included)
* history of gastric surgery
* emergency surgery such as perforation or obstruction
* other contraindication such as dysfunction of heart, lung, kidney

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Early gastric cancer patients with clinical stage T1N0M0
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The specificity of the Nomogram combining sentinel lymph node in predicting lymph node metastasis in early gastric cancer patients | 10 days after surgery when postoperative pathology result comes out

SECONDARY OUTCOMES:
The sensitivity of the Nomogram combining sentinel lymph node in predicting lymph node metastasis in early gastric cancer patients | 10 days after surgery when postoperative pathology result comes out
The sensitivity of the Nomogram alone in predicting lymph node metastasis in early gastric cancer patients | 10 days after surgery when postoperative pathology result comes out

CONTACTS AND LOCATIONS:
Overall Officials: Zhaode Bu, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China